CLINICAL TRIAL: NCT01847716
Title: Transforming Growth Factor Beta Signalling in the Development of Muscle Weakness in Pulmonary Arterial Hypertension
Status: Terminated | Type: Observational
Why Stopped: numbers recruited to show adequate association but not primary outcome
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council (Other Government); Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 13IC0457
Record Dates: First submitted 2013-04-19; First posted 2013-05-07 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Muscle Weakness; Pulmonary Arterial Hypertension
Keywords: Muscle weakness; Pulmonary arterial hypertension; Transforming growth factor beta; Growth and differentiation factor 15
MeSH Terms: conditions — Muscle Weakness; Pulmonary Arterial Hypertension; Camurati-Engelmann Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Muscle biopsy and blood specimens will be retained by Imperial College and are subject to thier restrictions ad regulations
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- PH with wasting: This group of patients with idiopathic pulmonary arterial hypertension exhibit quadriceps wasting
- PH no wasting: This groups of patients with idiopathic pulmonary arterial hypertension exhibit no evidence of muscle wasting
- Controls: This group of volunteers does not have pulmonary arterial hypertension and would not be expected to have muscle wasting

SUMMARY:
Pulmonary arterial hypertension (PAH) is a disease that causes raised blood pressure in blood vessels that pick up oxygen from the lungs. It has a life expectancy similar to some cancers. There is treatment available but there is no cure. We now know that PAH is associated with weakness in the muscles in the legs, which contributes to the symptoms patients' experience. Researchers believe that certain proteins found in high levels in the blood of patients with other chronic diseases can affect muscle function and growth. One of these proteins is called growth differentiating factor (GDF) 8, high levels of which are associated with muscle weakness in chronic obstructive pulmonary disease(COPD) and heart failure (HF). Interestingly there are drugs available which block the actions of GDF-8 on muscle cells which has been shown in animals to result in increased muscle size. A related protein called GDF-15 is found in elevated levels in patients PAH, and is linked to prognosis. Our preliminary data suggests that GDF-15 can also directly influence muscle size in a number of situations. We aim to investigate the role of GDF-15 and related molecules in the development of muscle weakness in patients with PAH. We will do this by measuring certain markers of muscle weakness and taking blood and muscle samples in patients and controls. We will then compare the levels of GDF-15 in these tissues in those with and without muscle wasting. We hope this work will lead to a greater understanding of the role of GDF-15 in the development of muscle weakness in patients with PAH. GDF-15 levels may be important in allowing us to define which patients have muscle weakness. In the future we aim to perform a clinical trial of drugs which block the actions of GDF-15.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pulmonary arterial hypertension with New York Heart Association stage II - III disease will be eligible for recruitment in the patient portion of the trial. Interested healthy age matched volunteers will also be recruited.

Exclusion Criteria:

* Patients and volunteers will be excluded if they have significant co-morbidities including other cardiorespiratory disease, metabolic abnormalities including diabetes or thyroid disorders. They will be excluded if they cannot safely exercise and perform a six minute walk test or if they are wheelchair bound.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinics at Royal Brompton and Hammersmith hospital
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2013-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Plasma growth and differentiation factor 15 levels in participants with and without muscle wasting | 30 months
  Muscle wasting will be defined by quadriceps cross sectional area measured by ultrasound

SECONDARY OUTCOMES:
Correlation of plasma Growth and differentiation factor 15 levels with muscle strength | 30 months
  Muscle strength will be measured by quadriceps maximal volitional capacity percent predicted
Change in fibre type in muscle biopsy | 30 months
GDF-15 levels in biopsy specimens | 30 months
Correlation of plasma Growth and differentiation factor 15 levels with brain natriuretic protein levels | 30 months
Correlation of plasma Growth and differentiation factor 15 levels with fat free mass index | 30 months
  Fat free mass index will be measured by bioelectrical impedence
Correlation of plasma Growth and differentiation factor 15 levels with quality of life | 30 months
  Quality of life will be measured by St. George's respiratory questionnaire
Correlation of plasma Growth and differentiation factor 15 levels with exercise tolerance | 30 months
  Exercise tolerance will be measured by six minute walk test
Correlation of plasma Growth and differentiation factor levels 15 with physical activity levels | 30 months
  Physical activity will be measured by Sensewear armband
Correlation of plasma Growth and differentiation factor levels 15 with echocardiographic measures of severity of pulmonary hypertension | 30 months
Correlation of GDF-15 levels in biopsy specimens with muscle wasting and weakness | 30 months
  Wasting will be measured by quadriceps cross sectional area and weakness will be defined by quadriceps maximal volitional capacity
Determine the contribution of atrophy and autophagy to muscle wasting in PAH | 30 months
  Muscle biopsy specimens will be evaluated using microscopy and real time polymerase chain reaction
Determine the contribution of SMAD and non-SMAD signalling pathways to the development of muscle weakness and wasting in PAH | 30 months
  Phosphorylation of SMAD and non-SMAD signalling will be determined by western blot

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Wort, MBBS, Principal Investigator — Imperial College / Royal Brompton Hospital
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Garfield BE, Crosby A, Shao D, Yang P, Read C, Sawiak S, Moore S, Parfitt L, Harries C, Rice M, Paul R, Ormiston ML, Morrell NW, Polkey MI, Wort SJ, Kemp PR. Growth/differentiation factor 15 causes TGFbeta-activated kinase 1-dependent muscle atrophy in pulmonary arterial hypertension. Thorax. 2019 Feb;74(2):164-176. doi: 10.1136/thoraxjnl-2017-211440. Epub 2018 Dec 15. PMID 30554141